CLINICAL TRIAL: NCT02943096
Title: Flavanol Augmentation for Antidepressant Non-Responsive Late Life Depression
Acronym: Flavanol
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study stopped due to funding limitations
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Columbia University (Other)
Responsible Party: Principal Investigator, Bret Rutherford, Associate Professor of Clinical Psychiatry, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7368
Record Dates: First submitted 2016-10-18; First posted 2016-10-24 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Depression; Major Depressive Disorder
MeSH Terms: conditions — Depression; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flavanol (Active Comparator): Blinded treatment with either CocoaVia 500mg or placebo.
  Interventions: Dietary Supplement: CocoaVia
- Placebo (Placebo Comparator): Blinded treatment with either CocoaVia 500mg or placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: CocoaVia — Flavanols represent a specific group of plant derived nutrients that are found in cocoa beans, grapes, tea, berries and various other fruits and vegetables. The specific flavanols investigated in this study come from cocoa.
  Arms: Flavanol
Other: Placebo — The placebo looks like the other intervention pills, but does not contain any flavanols (it is sometimes called a "sugar pill").
  Arms: Placebo

SUMMARY:
The goal of this proposal is to conduct the first pilot study of whether consuming flavanol supplements will augment the cognitive and mood benefits of antidepressant medication in older adults with Late LifeDepression (LLD). Flavanols represent a specific group of plant derived nutrients that are found in cocoa beans, grapes, tea, berries and various other fruits and vegetables. The specific flavanols investigated in this study come from cocoa. Currently available treatments for LLD (i.e., antidepressant medication) are limited in efficacy, especially in individuals who also suffer from cognitive impairment. Recent studies performed at Columbia and elsewhere suggest that flavanols may induce beneficial brain changes that support cognitive functioning and elevate mood, but their precise clinical effects in older adults with combined depression and cognitive impairment remain to be evaluated. For this study, the investigators plan to recruit 50 adults aged ≥60 years who have Major Depressive Disorder, meet a minimum depressive symptom threshold despite currently receiving an adequate trial of an antidepressant, and have a significant cognitive complaints without a diagnosis of dementia. Subjects will be randomized to receive 8 weeks of augmentation treatment with flavanol capsules (in addition to continuing their antidepressant) vs. capsules not containing flavanols. Pre- and post-treatment MRI scanning of the brain will be conducted, and comprehensive pre- and post-treatment neuropsychological assessment will be performed. Results from this project will allow the investigators to evaluate a novel therapeutic approach to LLD, which could have large public health ramifications given the prevalence, frequent treatment resistance, and chronicity characteristic of LLD.

DETAILED DESCRIPTION:
The goal of this proposal is to conduct the first pilot study of whether consuming a diet high in flavanols will augment the cognitive and mood benefits of antidepressant medication in older adults with Late Life Depression (LLD). LLD affects 3% of community-dwelling adults over 60 years old, and 15% of older adults living in the community have clinically significant depressive symptoms. Diagnosis with LLD increases an older adult's risk of disability by 67-73% over 6 year follow up, causes twice the functional impairment compared to those without LLD, and is associated with high rates of completed suicide in individuals over 65. Currently available treatments for LLD (i.e., antidepressant medication) are limited in efficacy, leading to high rates of recurrence and frequent development of chronicity. Cognitive impairment, which is commonly associated with LLD, predicts poor acute response to antidepressants, leads to higher relapse rates during the continuation phase of treatment, and is associated with the development of adverse age-related health outcomes, including increased risk of dementia, dependence in activities of daily living (ADL), and driving cessation.

Novel treatments addressing LLD's underlying neurobiology are critically needed, particularly therapies that may also have beneficial effects on the cognitive components of LLD. The most extensively studied brain region to be implicated in both the depressive and cognitive aspects of LLD has been the hippocampus. Decreased hippocampal volumes are found in depressed patients compared to controls, and this finding appears to be particularly pronounced in individuals with recurrent depressive illness. Among the subregions comprising the hippocampus, evidence suggests that it is decreased neurogenesis within the dentate gyrus (DG) specifically that may contribute to the development of depression, and it appears that part of the mechanism of action of antidepressants is to enhance neurogenesis in the DG. As the DG is also a critical contributor to the cognitive functions of the hippocampus, it stands out as a highly significant brain region that may be involved with both the mood and cognitive components of LLD.

ELIGIBILITY:
Inclusion Criteria

* Men and women aged ≥60 years (Method of ascertainment: clinical interview)
* DSM 5 diagnosis of Major Depressive Disorder (Method of ascertainment: SCID, clinical interview)
* Subjective report of memory or thinking problems (Method of ascertainment: clinical interview)
* 24-item Hamilton Rating Scale for Depression ≥16 (Method of ascertainment: HRSD)
* Failure of depressive symptoms to remit following an adequate trial of an antidepressant (defined as at least 8 weeks of treatment, with 4 weeks of at least half PDR maximum dose, of an FDA approved antidepressant) (Method of ascertainment: clinical interview)
* Capable of providing informed consent and complying with the study procedures (Method of ascertainment: clinical interview)

Exclusion Criteria

* Diagnosis of Substance Use Disorder within the past 12 months (excluding Tobacco) (Method of ascertainment: SCID, clinical interview)
* History of psychosis, psychotic disorder, mania, or bipolar disorder (Method of ascertainment: SCID, clinical interview)
* HRSD suicide item > 2 or CGI =7 at baseline (Method of ascertainment: HRSD, CGI)
* Diagnosis of probable or definite dementia (Alzheimer's Disease, Vascular Dementia, Parkinson's disease, etc.) (Method of ascertainment: SCID, clinical interview, MMSE)
* MMSE ≤24 (Method of ascertainment: MMSE)
* Physical or intellectual disability adversely affecting ability to complete assessments (Method of ascertainment: clinical interview)
* History of allergy, hypersensitivity, or intolerance to cocoa flavanols (Method of ascertainment: clinical interview)
* Contraindication to MRI scanning or unable to tolerate scanning procedures (Method of ascertainment: clinical interview)
* Allergic or adverse reaction to gadolinium, 2 or more prior scans with gadolinium, or creatinine clearance < 50 (Method of ascertainment: clinical interview, blood draw)
* Daily consumers of dietary or herbal supplements, including Gingko, flavonoid, and dietary herbal or plant extracts (Method of ascertainment: clinical interview)
* Diabetes or acute, severe, or unstable medical or neurologic condition (Method of ascertainment: clinical interview, physical exam, EKG)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-02-06 (Actual); Study Completion 2018-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bret Rutherford, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We will recruit subjects via advertisements for patients who feel depressed, through the RecruitMe online platform, as well as clinical referrals from colleagues around CUMC.
Pre-assignment Details: Every subject evaluated for this protocol will receive a clinical interview by a psychiatrist or psychologist, be administered the 24-item Hamilton Rating Scale for Depression (HRSD) and Antidepressant Treatment History Form, and have a SCID performed by a trained rater. They will be educated about appropriate treatments available for depression.
Period: Overall Study
Arm/Group | Flavanol | Placebo
Started | 3 | 3
Completed | 3 | 2
Not Completed | 0 | 1
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Flavanol | Placebo | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 2 | 3 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.8 (5.72) | 75.2 (8.93) | 73.5 (6.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 1 | 3 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6
Hamilton Rating Scale for Depression [Mean (Standard Deviation); unit: units on a scale] — Scale for depressive symptoms administered by trained rater. The HRSD is the standard measure of depression severity for clinical trials of antidepressants and was chosen as the primary outcome measure over other depression rating scales to ensure compatibility of study results with our meta-analyses and ongoing studies of expectancy. Although the HRSD list 21 items, the scoring is based on the first 24 items. The minimum score is 0 and the maximum score is 74. The higher the number the worse outcome.
  units on a scale | 20 (1.73) | 17 (8.72) | 18.5 (5.86)

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Rating Scale of Depression (HRSD)
Description: Scale for depressive symptoms administered by trained rater. The HRSD is the standard measure of depression severity for clinical trials of antidepressants and was chosen as the primary outcome measure over other depression rating scales to ensure compatibility of study results with our meta-analyses and ongoing studies of expectancy. Although the HRSD list 21 items, the scoring is based on the first 24 items. The minimum score is 0 and the maximum score is 74. The higher the number the worse outcome.
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Flavanol | Placebo
Number analyzed (Participants) | 3 | 3
score on a scale | 18.3 (6.43) | 20.3 (2.08)

2. Secondary Outcome: Mnemonic Similarity Task (MST)
Description: First, participants had to complete an encoding task were they were shown 128 items, ½ objects(2 seconds) and ½ scene (3 seconds). Right after, they were given instructions on a video on how to do the test phase. They were instructed to identified the following images as "old", "similar", or "new". They were then shown 192 items: 64 old items, 64 lures (similar), and 64 foil (new) for 2.5 seconds (objects)/3 seconds (scene). The images were intermixed during the test. The Lure Discrimination Index was calculated as the difference between the rate of "similar" responses give to lure items minus "similar" responses given to foil. This corrected for response bias. Correct responses are those that were identified correctly by the participant. A negative response means that the number of answered correctly was less that those answered incorrectly.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Percent Endorsed
Arm/Group | Flavanol | Placebo
Number analyzed (Participants) | 3 | 3
Percent Endorsed | -0.0567 (.031) | 0.28 (0.178)

3. Secondary Outcome: Modified-Benton Task (ModBent)
Description: The ModBent assesses pattern separation, a measure of cognitive functioning. The task was created to measure dentate gyrus-dependent cognition. It shows participants patterns for 10 seconds, then presents two patterns afterwards on a different screen. Participants are then asked to determine which of the two patterns is the one they previously studied for 10 seconds. The second component of the task then goes through a series of patterns, one by one - the participant has to then decide whether each pattern was one they previously studied for 10 seconds or not. We analyzed the mean Reaction time for correct rejections.
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: millisecond
Arm/Group | Flavanol | Placebo
Number analyzed (Participants) | 3 | 3
millisecond | 5459.22 (592.67) | 5820.29 (675.79)

4. Secondary Outcome: Modified-Benton Task (ModBent)
Description: as for outcome 3
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: millisecond
Arm/Group | Flavanol | Placebo
Number analyzed (Participants) | 3 | 3
millisecond | 4081.04 (412.17) | 6000.02 (403.67)

5. Secondary Outcome: Mnemonic Similarity Task (MST)
Description: as for outcome 2
Time Frame: Week 8
Measure: Median (Standard Deviation); unit: Percent Endorsed
Arm/Group | Flavanol | Placebo
Number analyzed (Participants) | 3 | 3
Percent Endorsed | 0.15 (0.32) | .61 (0.29)

ADVERSE EVENTS:
Time Frame: 8 Weeks
Arm/Group | Flavanol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-08-30): https://cdn.clinicaltrials.gov/large-docs/96/NCT02943096/Prot_SAP_ICF_000.pdf